CLINICAL TRIAL: NCT01374152
Title: A Randomized Controlled Trial of Cognitive Sensory Motor Training Therapy on the Recovery of Upper Extremity Function in Acute Stroke Patients
Brief Title: Perfetti Method in Upper Extremity of Stroke Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prasat Neurological Institute (Other Government)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Ratanapat Chanubol, Dr., Prasat Neurological Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Perfetti
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Stroke
Keywords: stroke; upper extremity; rehabilitation; perfetti
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perfetti (Experimental): Cognitive sensory motor training method for upper extremities rehabilitation every working day, totally training not less than 600 minutes within 4 weeks.
  Interventions: Other: cognitive sensory motor training therapy
- conventional rehabilitation (No Intervention): conventional occupational therapy method for upper extremities rehabilitation every working day, totally training not less than 600 minutes within 4 weeks.

INTERVENTIONS:
Other: cognitive sensory motor training therapy — training method that emphasis on cognition/ sensation/ and motor movement together train every working day 45 minutes per day for 4 weeks.
  Other Names: Perfetti; Cognitive sensory motor training; Stroke; Upper extremity
  Arms: Perfetti

SUMMARY:
The cognitive sensory motor training therapy (Perfetti's technique) might be more effectiveness than conventional occupational therapy on upper extremity function recovery after acute stroke patients.

DETAILED DESCRIPTION:
Globally, stroke is the second leading cause of death above the age of 60 years, and the fifth leading cause of death in people aged 15 to 59 years old. Upper extremities problem is still faced with poor prognosis for recovery. Cognitive sensory motor training therapy (Perfetti's technique) might be better helped for recovery of upper extremity function in stroke than conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* First ever stroke
* Impaired upper extremity function
* Given signed inform consent

Exclusion Criteria:

* Unstable medical condition
* Any upper extremity functional impairment prior to stroke
* Can not adequately cooperate in training
* Severe communication problems
* Severe cognitive - perceptual deficits
* Fixed contracture more than 30 degree in every upper extremity joint

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Action research arm test | 4 weeks
  The Action research arm test used for assess the impairment of upper limb function. ARAT has ordinal 4-point scale (0-3) in 19 items. Totally 57 scores.

SECONDARY OUTCOMES:
Box and block test | 4 weeks.
  For evaluated gross manual dexterity, consist of two adjacent boxes of the same size. Between the two boxes, there is a partition. It is recorded the number of wooden block that can be transported from one compartment of a box to another within 60 seconds
Extended Barthel Index | 4 weeks.
  Basic activity of daily living and degree of independence from any form of help.

CONTACTS AND LOCATIONS:
Overall Officials: Ratanapat Chanubol, MD., Principal Investigator — Prasat Neurological Institute
Locations (1):
- Prasat neurological institute, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Wongphaet P, Butrach W, Sangkrai S, Jitpraphai C. Improved function of hemiplegic upper extremity after cognitive sensory motor training therapy in chronic stroke patients: preliminary report of a case series. J Med Assoc Thai. 2003 Jun;86(6):579-84. PMID 12924807
- [Background] Duncan PW, Goldstein LB, Horner RD, Landsman PB, Samsa GP, Matchar DB. Similar motor recovery of upper and lower extremities after stroke. Stroke. 1994 Jun;25(6):1181-8. doi: 10.1161/01.str.25.6.1181. PMID 8202977
- [Background] Lyle RC. A performance test for assessment of upper limb function in physical rehabilitation treatment and research. Int J Rehabil Res. 1981;4(4):483-92. doi: 10.1097/00004356-198112000-00001. No abstract available. PMID 7333761